CLINICAL TRIAL: NCT01162928
Title: Assessment of the Benefit From Combined Administration of Oral and Intravenous Nutrition - Enriched With Omega-3 Fatty Acids - for Intensive Care Patient
Brief Title: Parenteral Nutrition With Intravenous and Oral Fish Oil for Intensive Care Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-0804; NCT01148589 (obsolete NCT alias)
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness
Keywords: critically ill, mechanically ventilated patients requiring enteral and parenteral nutritional support
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 3-chamber-bag combined with Oxepa
  Interventions: Drug: Nutriflex Omega special + Oxepa
- 2 (Active Comparator): 3-chamber-bag combined with Pulmocare
  Interventions: Drug: Nutriflex Lipid special + Pulmocare

INTERVENTIONS:
Drug: Nutriflex Omega special + Oxepa — 3-chamber-bag combined with enteral nutrition
  Arms: 1
Drug: Nutriflex Lipid special + Pulmocare — 3-chamber-bag combined with enteral nutrition
  Arms: 2

SUMMARY:
The primary objective is to assess the effect of fish oil-enriched enteral and parenteral nutrition on blood oxygenation in critically ill patients.

ELIGIBILITY:
Inclusion: - signed informed consent

* mechanically-ventilated adults (age 18-80) admitted to Intensive Care Unit,
* enteral nutrition does not meet the nutrition goal (at least 80 % of the resting energy expenditure) within the past 36 hours
* APACHE II score above the median value of the intensive care unit (id est > 20)

Exclusion: - do not resuscitate status

* cardiogenic pulmonary edema
* previous (< 1 month) or ongoing need for corticosteroids > 0.1 mg/kg prednisolon- equi-valent or other immune suppressive treatment
* serum triglycerides > 300 mg/dl at screening
* alterations of coagulation (platelets <100.000 mm3), PTT > 60 sec, INR ≥ 2.5 without therapeutic intervention
* pregnancy
* participation in a clinical study with an investigational drug within one month prior to the start of this clinical trial
* known or suspected drug abuse
* general contraindications for infusion therapy such as acute pulmonary oedema, hyper-hydration and decompensated cardiac insufficiency
* known hypersensitivity to egg-, soy-, and fish proteins or any of the ingredients
* autoimmune disease or HIV
* uncompensated hemodynamical failure of any origin (hemorrhagic shock, myocardial infarction, cardiac failure)
* uncompensated ketoacidosis caused by Diabetes mellitus within 7 days prior to onset of study
* uncompensated renal insufficiency with serum creatinine > 1.5 mg/dL (> 133 µmol/L)
* patients with severe liver dysfunction with bilirubin > 2.5 mg/dL (> 43 µmol/L)
* necrotizing pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
change in blood oxygenation (PaO2/FIO2 ratio) | day 1 to day 6

SECONDARY OUTCOMES:
rate of parenteral nutrition associated complications equal or better compared to current practice | day 1 to day 6
disease related complications | Day 28
28 day-mortality | Day 28
changes in fatty acid composition of cell membranes | Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, MD, Principal Investigator — Rabin Medical Center, Beilinson Campus
Locations (1):
- Rabin Medical Center, Beilinson Campus, Petah Tikva, Israel

REFERENCES:
- [Derived] Singer P, Bendavid I, Mesilati-Stahy R, Green P, Rigler M, Lev S, Schif-Zuck S, Amiram A, Theilla M, Kagan I. Enteral and supplemental parenteral nutrition enriched with omega-3 polyunsaturated fatty acids in intensive care patients - A randomized, controlled, double-blind clinical trial. Clin Nutr. 2021 May;40(5):2544-2554. doi: 10.1016/j.clnu.2021.03.034. Epub 2021 Apr 1. PMID 33932802